CLINICAL TRIAL: NCT04244162
Title: Mechanisms Mediating Postoperative Neurocognitive Disorders
Brief Title: Postoperative Neurocognitive Disorders
Acronym: PNCD
Status: Completed | Type: Observational
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Susana Vacas, MD, PhD, Physician, Massachusetts General Hospital
Other Study IDs: PNCD 19-001597
Record Dates: First submitted 2020-01-23; First posted 2020-01-28 (Actual); Last update posted 2025-11-03 (Actual); Status verified 2025-10

CONDITIONS: Obstructive Sleep Apnea; Neurocognitive Disorders
Keywords: brain imaging; neurocognitive testing
MeSH Terms: conditions — Sleep Apnea, Obstructive; Neurocognitive Disorders | interventions — Neuroimaging

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Study Group: brain scans, cognitive tests, blood biomarkers
  Interventions: Diagnostic Test: Brain Imaging; Diagnostic Test: Cognitive testing; Diagnostic Test: Blood Biomarkers

INTERVENTIONS:
Diagnostic Test: Brain Imaging — Magnetic resonance imaging (MRI) using diffusion tensor imaging (DTI)-based mean diffusivity (MD) measures.
Diagnostic Test: Cognitive testing — Wide Range Assessment of Memory and Learning (WRAML2), Montreal Cognitive Assessment (MoCA), and Confusion Assessment Method for the ICU -severity (CAM-ICU S) tests.
Diagnostic Test: Blood Biomarkers — Inflammatory markers

SUMMARY:
The purpose of this study is to examine the mechanisms of brain injury contributing to postoperative neurocognitive disorders (PNCD) in an at-risk population (obstructive sleep apnea (OSA)) undergoing surgery. The investigators will enroll 50 OSA patients scheduled for surgery. All patients will have a brain scan (fMRI) within five days before surgery and two days and six months after surgery. During this visit cognitive function will be assessed using the Wide Range Assessment of Memory and Learning (WRAML2) and Montreal Cognitive Assessment (MoCA) tests. Patients will also be asked to participate in a blood draw during the first 2 visits for fMRI (within five days of surgery and two days after surgery). The Confusion Assessment Method (CAM-S) test, will be used to examine postoperative delirium.

DETAILED DESCRIPTION:
The investigators will examine the potential mechanisms of brain injury contributing to postoperative neurocognitive disorders (PNCD) in an at-risk population (obstructive sleep apnea (OSA)). This study proposes that neuro-inflammation is associated with measurable tissue changes that can be examined with MD measures and blood biomarkers.

On the day of surgery, standard of care procedures will take place. Hemodynamic vitals will be continuously monitored. As per the latest guidelines and recommendations from the American Society of Anesthesiologists (ASA), mean arterial pressure (MAP) will be targeted to > 60 mmHg or within 20% of baseline values, and processed EEG-guided anesthesia will be monitored to maintain a patient state index between 20-50. Electronic medical records and intraoperative integrated physiologic waveform will be collected.

In summary, the investigators will examine the potential mechanisms of brain injury contributing to postoperative delirium (POD) and acute and long-lasting neurocognitive deficits in an at-risk population (OSA).

ELIGIBILITY:
Inclusion Criteria:

Subjects with a diagnosis of moderate-to-severe OSA (apnea hypopnea index [AHI]>15 events/hour confirmed by overnight polysomnography), scheduled for open or robotic surgery (abdominal, gynecologic, or urologic), and upper or lower extremity orthopedic procedures

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects with a diagnosis of moderate-to-severe OSA (apnea hypopnea index [AHI]>15 events/hour confirmed by overnight polysomnography),
Sampling Method: Non-Probability Sample
Enrollment: 32 (Actual)
Dates: Start 2020-12-12 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2025-08-31 (Actual)

PRIMARY OUTCOMES:
Preoperative cognitive function | pre-surgery (within five days before)
  Montreal Cognitive Assessment (MoCA) test
Postoperative cognitive dysfunction - delayed cognitive recovery | Post-surgery (within two days post surgery).
  Montreal Cognitive Assessment (MoCA) test
Postoperative cognitive dysfunction - neurocognitive disorder | Post-surgery (6 months after surgery).
  Montreal Cognitive Assessment (MoCA) test
Preoperative cognitive function II | pre-surgery (within five days before surgery)
  Wide Range Assessment of Memory and Learning (WRAML2)
Postoperative cognitive dysfunction - delayed cognitive recovery II | Post-surgery (within two days post surgery).
  Wide Range Assessment of Memory and Learning (WRAML2)
Postoperative cognitive dysfunction - neurocognitive disorder II | Post-surgery (6 months after surgery).
  Wide Range Assessment of Memory and Learning (WRAML2)
Postoperative Delirium | A two times per day for up to three days or discharge from the hospital.
  The Confusion Assessment Method (CAM-S) test

SECONDARY OUTCOMES:
Blood Serum anti-inflammatory Biomarkers | pre- (within five days before surgery)
  Assess blood inflammatory biomarkers (IL6, TNFa and IL1B) using enzyme-linked immunosorbent assay
Blood Serum anti-inflammatory Biomarkers II | post-surgery (within two days of surgery).
  Assess blood inflammatory biomarkers (IL6, TNFa and IL1B) using enzyme-linked immunosorbent assay
Brain changes | pre- (within five days before) and post-surgery (within two days and 6 months).
  Using non-invasive magnetic resonance imaging based diffusion tensor imaging
Brain changes II | Post-surgery (within two days post surgery).
  Using non-invasive magnetic resonance imaging based diffusion tensor imaging
Brain changes III | Post-surgery (within six months post surgery).
  Using non-invasive magnetic resonance imaging based diffusion tensor imaging

CONTACTS AND LOCATIONS:
Overall Officials: Rajesh Kumar, PhD, Principal Investigator — University of California, Los Angeles
Locations (1):
- Ronald Reagan UCLA Medical Center, Department of Anesthesiology & Perioperative Medicine, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No